CLINICAL TRIAL: NCT00495261
Title: Development and Validation of a Mindfulness Intervention for Problem Gambling: An Exploratory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Tony Toneatto, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 311/2006
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Gambling
Keywords: Gambling; Mindfulness; Cognitive Behavioural Therapy
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Mindfulness-enhanced cognitive behavioural therapy (MCBT)
- 2 (Active Comparator)
  Interventions: Behavioral: relaxation-enhanced cognitive behavioural therapy (RCBT)

INTERVENTIONS:
Behavioral: Mindfulness-enhanced cognitive behavioural therapy (MCBT) — a variation of cognitive behavioural therapy (CBT)
  Arms: 1
Behavioral: relaxation-enhanced cognitive behavioural therapy (RCBT) — a variation of cognitive behavioural therapy (CBT)
  Arms: 2

SUMMARY:
In recent years, mindfulness meditation has been shown to be a promising approach for alleviating emotional distress associated with chronic medical and psychiatric conditions and in reducing relapse following treatment for depression. The applicability of mindfulness meditation to problem gambling has not yet been explored. Mindfulness meditation may be particularly suitable for this clinical disorder as it stresses a process-oriented, metacognitive, approach to cognitive pathology in contrast to a content-focused approach, characteristic of traditional approaches to treating cognitive psychopathology. Gambling-related cognitive psychopathology is a well-known characteristic of problem gambling and frequently the target of therapy. Although there is growing evidence that cognitive-behavioral treatments are effective for gambling, outcomes may be improved by teaching gamblers additional ways to cope with cognitive distortions that emphasize metacognitive processes.

DETAILED DESCRIPTION:
Hypothesis The mindfulness-enhanced CBT (MCBT) will report significant reductions in the frequency of gambling, gambling urges, gambling cognitions and gambling-related expenditures compared to the relaxation-enhanced CBT (RCBT) at end-of-treatment and at the 3-month follow-up.

Significance

1. feasibility of mindfulness interventions for problem gamblers
2. tentative data for the effectiveness of the intervention
3. an additional clinical tool to treat problem gamblers
4. basis of a larger, grant-funded study obtain more definitive data

ELIGIBILITY:
Inclusion Criteria:

* current diagnosis of pathological gambling
* willingness to practice mindfulness or relaxation

Exclusion Criteria:

* substance abuse/dependence (except nicotine)
* concurrent attendance at any treatment in which their gambling is addressed (including Gamblers Anonymous)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Gambling urges | Baseline, post and 3 month fup
Gambling-related expenditures | Baseline, post and 3 month fup

SECONDARY OUTCOMES:
treatment adherence | Baseline, post and 3 month fup
gambling cognitions | Baseline, post and 3 month fup

CONTACTS AND LOCATIONS:
Overall Officials: Tony Toneatto, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada